CLINICAL TRIAL: NCT05087290
Title: Longer-term Effects of COVID-19 on Blood Vessels and Blood Pressure (LOCHINVAR) Phenotyping Study
Brief Title: LOnger-term Effects of COVID-19 INfection on Blood Vessels And Blood pRessure (LOCHINVAR)
Acronym: LOCHINVAR
Status: Completed | Type: Observational
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Sandosh Padmanabhan, Professor Sandosh Padmanabhan, University of Glasgow
Other Study IDs: GN20CA501; 21/WS/0075 (Other: NHS Greater Glasgow and Clyde); 299056 (Other: IRAS); RG2690/21/24 (Other Grant/Funding Number: HEART Research UK)
Record Dates: First submitted 2021-10-18; First posted 2021-10-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hypertension; Covid19
Keywords: Hypertension; COVID-19
MeSH Terms: conditions — Hypertension; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — With consent from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: SARS-CoV-2 +ve cases
  Interventions: Other: Cases
- Control: SARS-CoV-2 -ve cases
  Interventions: Other: Controls

INTERVENTIONS:
Other: Cases — All performed at baseline, 12 months and 18 months Medical and drug history Anthropometric tests Electrocardiogram Brachial flow mediated dilatation 6 minute walk test Blood sampling Urine sampling 24-hr Ambulatory Blood Pressure Monitor Questionnaires
  Optional:
  Stool sampling,24-hr Urine collection, Home Blood Pressure Monitor
  Groups: Cases
Other: Controls — All performed at baseline, 12 months and 18 months Medical and drug history Anthropometric tests Electrocardiogram Brachial flow mediated dilatation 6 minute walk test Blood sampling Urine sampling 24-hr Ambulatory Blood Pressure Monitor Questionnaires
  Optional:
  Stool sampling,24-hr Urine collection, Home Blood Pressure Monitor
  Groups: Control

SUMMARY:
The COVID-19 pandemic is the biggest medical challenge in decades. Individuals with pre-existing cardiovascular diseases have a higher risk of severe disease and death from COVID-19. The SARS-CoV-2 virus causes infection by targeting a molecule on the walls of the cells lining the lungs and the blood vessels leading to injury. There are concerns that after recovery from COVID-19, the damage sustained by these cells may have long-term consequences including high blood pressure, stroke and heart attacks. The burden of high blood pressure as a result of the pandemic is unknown and a greater understanding of COVID-19 impact on blood pressure and its underlying mechanisms is urgently needed.

LOCHINVAR is based on our pilot study "COVID-19 blood pressure endothelium interaction study" (OBELIX,NCT04409847, IRAS 284453), which found that patients with normal blood pressure at the time of hospital admission with COVID-19 showed a nine-point higher blood pressure ≥12 weeks after recovery, compared to a group without COVID-19. LOCHINVAR will extend the OBELIX study aiming to establish if COVID-19 increases the risk of developing high blood pressure and investigating underlying mechanisms through detailed measurements of blood pressure, blood vessel function, hormones and chemicals in the blood, urine and stool.

The investigators will invite 150 adults without pre-existing high blood pressure who were discharged from hospital after an admission: half with COVID-19 and half without. Baseline visit will be ≥12 weeks after discharge for measurements of blood pressure, tests of heart and blood vessel health, blood, urine and stool samples along with questionnaires on mood and quality of life. Two further study visits follow, at 12 and 18 months.

This study will generate crucial evidence on the long-term impact of COVID-19 on blood pressure along with information on potential mechanisms of this effect with immediate, transferable impact on clinical practice and inform risk mitigation measures.

DETAILED DESCRIPTION:
The Coronavirus Disease-19 (COVID-19) pandemic is one of the biggest medical challenges in recent years. Whilst COVID-19 primarily affects the lungs, causing interstitial pneumonitis and severe acute respiratory distress syndrome, it also affects multiple organ systems, including the cardiovascular system(1-3). There are documented associations between severity of disease/mortality risk and advancing age, male sex and associated comorbid disease (hypertension, ischaemic heart disease, diabetes, obesity, COPD and cancer).(4,5) The most common complications include cardiac dysrhythmia(6,7), cardiac injury(8,9), myocarditis, heart failure, pulmonary embolism10 and disseminated intravascular coagulation(11).

The SARS-CoV-2 virus uses the ACE2 receptor (ACE2) to enter type 2 pneumocytes, macrophages, perivascular pericytes, and cardiomyocytes.(12) This may lead to myocardial dysfunction and damage, endothelial dysfunction, microvascular dysfunction, plaque instability, and myocardial infarction.(12) In addition, ACE2 is expressed in several other organs including cells lining the blood vessels (endothelial cells), ACE2 is a key player in the renin-angiotensin system (RAS) which is important in blood pressure regulation and is a target for some of the commonly used drugs used in the treatment of blood pressure. While ACE2 is essential for viral invasion, it is unclear if the use of the common antihypertensive drugs ACE inhibitors or angiotensin receptor blockers (ARBs) alter prognosis in those with COVID-19 infection.(12) Furthermore, there is evidence that the normally occurring bacteria in the gut (gut microbiome) directly influences the makeup of the human immune system and has been implicated in severity of COVID-19 as well as in the magnitude of the immune system response to SARS-CoV-2 infection(13).

This study (LOCHINVAR) is based on the pilot study "COVID-19 blood pressure endothelium interaction study" (OBELIX), funded by the Chief Scientific Office. Preliminary results showed that participants who had COVID-19 infection had an 8.6mmHg increase in their average 24hr systolic blood pressure, compared to those that did not have COVID-19 infection. The investigators will increase our recruitment of potential participants to meet our sample size of 150 participants (75 SARS-CoV-2 +ve cases and 75 SARS-CoV-2 -ve cases) built on OBELIX. This study will allow us to have a better understanding of the risks of developing high blood pressure or uncontrolled blood pressure following COVID-19 infection. This will allow doctors to be able to make a recommendation on the current/long term management of people with high blood pressure beyond the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60 years
* Admission between 01/09/2020 - 31/12/2021
* Clinically suspected or Confirmed COVID-19 Reverse Transcription-Polymerase Chain Reaction (RT-PCR) test confirmed COVID-19 on admission
* No history of hypertension or current drug treatment for hypertension

Controls

1. Age 30-60
2. No history of hypertension
3. No antihypertensive drugs
4. Confirmed RT-PCR test negative and admission through Queen Elizabeth University Hospital immediate assessment unit and acute receiving units 01/09/2020 to 31/12/2021 or no history of SARS-CoV-2 infection or COVID-19

Exclusion Criteria:

Inability to give informed consent/lack of capacity BMI >40 eGFR <60 ml/min Pregnancy History of

* Cancer within 5 years
* Persistent atrial fibrillation
* Severe illness, at investigator discretion Prescription of
* BP lowering drugs
* Oral Corticosteroid (chronic use)
* Immunosuppressive agents
* Oral NSAIDs (chronic use)

Ages: 30 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients admitted through Queen Elizabeth University Hospital (QEUH) receiving units with suspected/confirmed COVID-19 during 01/09/2020-31/12/2021 and who are alive at discharge. Clinically suspected COVID-19 should have either fever, new onset cough and/or anosmia/dysgeusia and/or ≥2 of the following presenting features (fatigue/generalised weakness, headache, myalgia, sore throat/coryzal symptoms, breathlessness, anorexia/nausea/vomiting, diarrhoea, contact with known COVID-19 positive case). OBELIX participants who have given consent previously will be re-contacted.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
24-hour ABPM Systolic Blood Pressure | 12 months
  Average 24 hour Ambulatory Blood Pressure Monitoring - Systolic Blood Pressure , (all day and night) at 12 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls

SECONDARY OUTCOMES:
24-hour ABPM Diastolic Blood Pressure | 12 months and 18 months
  Average 24 hour Ambulatory Blood Pressure Monitoring - Diastolic Blood Pressure, 24hr (all day and night) at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Day ABPM Systolic Blood Pressure | 12 months and 18 months
  Day Ambulatory Blood Pressure Monitoring (Average Systolic Blood Pressure) 8 am to 8 pm at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Day ABPM Diastolic Blood Pressure | 12 months and 18 months
  Day Ambulatory Blood Pressure Monitoring (Average Diastolic Blood Pressure), 8 am to 8 pm at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Night ABPM Systolic Blood Pressure | 12 months and 18 months
  Night Ambulatory Blood Pressure Monitoring (Average Systolic Blood Pressure) 8pm to 8 am at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Night ABPM Diastolic Blood Pressure | 12 months and 18 months
  Night Ambulatory Blood Pressure Monitoring (Average Diastolic Blood Pressure) 8pm to 8 am at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
24-hour ABPM Heart Rate | 12 months and 18 months
  24 hour Ambulatory Blood Pressure Monitoring - Heart Rate, 24hr (all day and night) at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
24-hour Urine Sodium | 12 months and 18 months
  24-hour Urine Sodium at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls

OTHER OUTCOMES:
% Flow Mediated Dilatation | 12 months and 18 months
  % Brachial Flow Mediated Dilatation at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Exercise tolerance - distance walked in 6 minutes | 12 months and 18 months
  Exercise tolerance distance walked in 6 minutes at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Quality of life and mood - difference in longitudinal changes in QoL and mood between groups | 12 months and 18 months
  Patient Health Questionaire-9 (Minimal Depression 0-4, Mild Depression 5 - 9, Moderate Depression 10-14, Moderately Severe Depression 15 - 19, Severe Depression 20-27) and Euroqol (EQ5D-3L) Questionnaire (Mean EQ-5D and Standard Deviation) at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Mean Home Systolic Blood Pressure | 12 months and 18 months
  Mean Home Blood Pressure Measurements - Systolic Blood Pressure at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Mean Home Diastolic Blood Pressure | 12 months and 18 months
  Mean Home Blood Pressure Measurements - Diastolic Blood Pressure at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Day Home Systolic Blood Pressure | 12 months and 18 months
  Average Day Home Blood Pressure Measurements - Systolic Blood Pressure at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Evening Home Systolic Blood Pressure | 12 months and 18 months
  Average Evening Home Blood Pressure Measurements - Systolic Blood Pressure at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Day Home Diastolic Blood Pressure | 12 months and 18 months
  Average Day Home Blood Pressure Measurements - Diastolic Blood Pressure at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls
Evening Home Diastolic Blood Pressure | 12 months and 18 months
  Average Evening Home Blood Pressure Measurements - Diastolic Blood Pressure at 12 months and 18 months in SARS-CoV-2 +ve cases and in SARS-CoV-2 -ve controls

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Sandosh Padmanabhan, Glasgow, United Kingdom

REFERENCES:
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Driggin E, Madhavan MV, Bikdeli B, Chuich T, Laracy J, Biondi-Zoccai G, Brown TS, Der Nigoghossian C, Zidar DA, Haythe J, Brodie D, Beckman JA, Kirtane AJ, Stone GW, Krumholz HM, Parikh SA. Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the COVID-19 Pandemic. J Am Coll Cardiol. 2020 May 12;75(18):2352-2371. doi: 10.1016/j.jacc.2020.03.031. Epub 2020 Mar 19. PMID 32201335
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Liu K, Fang YY, Deng Y, Liu W, Wang MF, Ma JP, Xiao W, Wang YN, Zhong MH, Li CH, Li GC, Liu HG. Clinical characteristics of novel coronavirus cases in tertiary hospitals in Hubei Province. Chin Med J (Engl). 2020 May 5;133(9):1025-1031. doi: 10.1097/CM9.0000000000000744. PMID 32044814
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Lippi G, Lavie CJ, Sanchis-Gomar F. Cardiac troponin I in patients with coronavirus disease 2019 (COVID-19): Evidence from a meta-analysis. Prog Cardiovasc Dis. 2020 May-Jun;63(3):390-391. doi: 10.1016/j.pcad.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32169400
- [Background] Danzi GB, Loffi M, Galeazzi G, Gherbesi E. Acute pulmonary embolism and COVID-19 pneumonia: a random association? Eur Heart J. 2020 May 14;41(19):1858. doi: 10.1093/eurheartj/ehaa254. No abstract available. PMID 32227120
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Guzik TJ, Mohiddin SA, Dimarco A, Patel V, Savvatis K, Marelli-Berg FM, Madhur MS, Tomaszewski M, Maffia P, D'Acquisto F, Nicklin SA, Marian AJ, Nosalski R, Murray EC, Guzik B, Berry C, Touyz RM, Kreutz R, Wang DW, Bhella D, Sagliocco O, Crea F, Thomson EC, McInnes IB. COVID-19 and the cardiovascular system: implications for risk assessment, diagnosis, and treatment options. Cardiovasc Res. 2020 Aug 1;116(10):1666-1687. doi: 10.1093/cvr/cvaa106. PMID 32352535
- [Background] Segal JP, Mak JWY, Mullish BH, Alexander JL, Ng SC, Marchesi JR. The gut microbiome: an under-recognised contributor to the COVID-19 pandemic? Therap Adv Gastroenterol. 2020 Nov 24;13:1756284820974914. doi: 10.1177/1756284820974914. eCollection 2020. PMID 33281941
- [Derived] Lip S, Tran TQB, Hanna R, Nichol S, Guzik TJ, Delles C, McClure J, McCallum L, Touyz RM, Berry C, Padmanabhan S. Long-term effects of SARS-CoV-2 infection on blood vessels and blood pressure - LOCHINVAR. J Hypertens. 2025 Jun 1;43(6):1057-1065. doi: 10.1097/HJH.0000000000004013. Epub 2025 Apr 10. PMID 40178227
- [Derived] Lip S, Mccallum L, Delles C, McClure JD, Guzik T, Berry C, Touyz R, Padmanabhan S. Rationale and Design for the LOnger-term effects of SARS-CoV-2 INfection on blood Vessels And blood pRessure (LOCHINVAR): an observational phenotyping study. Open Heart. 2022 Jun;9(1):e002057. doi: 10.1136/openhrt-2022-002057. PMID 35750422
- See also: OBELIX Study — https://clinicaltrials.gov/ct2/show/NCT04409847?cond=COVID-19&cntry=GB&city=Glasgow&draw=2&rank=7